CLINICAL TRIAL: NCT06400693
Title: Evaluation and Comparison of Cognitive Aids in Emergency Airway Equipment Preparation: the Randomized, Controlled Template Airway Trial
Brief Title: Templates as Cognitive Aids in Emergency Airway Equipment Preparation: the Template Airway Trial
Acronym: TemplateAirway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Katharina Epp, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-17375
Record Dates: First submitted 2024-04-14; First posted 2024-05-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Airway Management
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Intervention Model Description: single-center, randomized, controlled simulation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Template (Other): Template is provided to prepare necessary equipment for emergency airway management
  Interventions: Other: Endotracheal Intubation; Other: Supraglottic Airway
- No template (Other): No template is provided to prepare necessary equipment for emergency airway management
  Interventions: Other: Endotracheal Intubation; Other: Supraglottic Airway

INTERVENTIONS:
Other: Endotracheal Intubation — Preparation of all necessary equipment for endotracheal intubation
Other: Supraglottic Airway — Preparation of all necessary equipment for laryngeal mask

SUMMARY:
Comparison of preparation times (in seconds) for emergency airway management (equipment only) with and without a template.

DETAILED DESCRIPTION:
Comparison of time (in seconds) needed to prepare all necessary equipment for one form of emergency airway management with and without a template. Participants will be randomized to "preparation with template (A)" and "preparation without template (B)" and all participants will be measured twice for both arms A and B, however, evaluation will take place on two separate days. Methods of airway management evaluated will be endotracheal intubation, supraglottic airway device and oral fiberoptic intubation, with a total of three measurements per participant per study day and two study days per participant. Participants will be nurses in the intensive care unit and, as a control group, anesthesia nurses will also be evaluated in order to factor in the effects of experience. The study will take place in the usual work environment of participants and with the standard equipment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* written informed consent
* Qualification as a nurse (ICU or anesthesia)
* employed with University Medical Centre of Johannes Gutenberg University (JGU) Mainz

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Time (in seconds) until completion of preparation of necessary equipment for endotracheal intubation between both groups | Defined verbal sign of participant when given task is started and ended
  Comparison of time (in seconds) until completion of preparation of necessary equipment for endotracheal intubation with and without template

SECONDARY OUTCOMES:
Time (in seconds) until completion of preparation of necessary equipment for supraglottic airway device between both groups | Defined verbal sign of participant when given task is started and ended
  Comparison of time (in seconds) until completion of preparation of necessary equipment for supraglottic airway device with and without template
Number of missing equipment for endotracheal intubation | immediately after completion of intervention
  Comparison of number of missing equipment for endotracheal intubation with and without template
Number of missing equipment for supraglottic airway between groups | immediately after completion of intervention
  Comparison of missing equipment for supraglottic airway with and without template
Number of wrong size/equipment between groups | immediately after completion of intervention
  Comparison of number of wrong size/equipment with and without template
Nasa Task Load Index | immediately after completion of all 3 assigned interventions on each study day
  Comparison of work load using Nasa Task Load Index questionnaire with and without template

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Epp, M.D., Principal Investigator — Employee
Locations (1):
- Department of Anaesthesiology, University Medical Centre of Johannes Gutenberg University, Mainz, Rhineland-Palatine, Germany

IPD SHARING:
Plan to Share IPD: No